CLINICAL TRIAL: NCT02955563
Title: CSDM: A Trial to Improve Communication and Shared Decision Making Using a Web-Based Tool
Acronym: CSDM Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Douglas White, Vice Chair and Professor of Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO16050247
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Intervention Compliance; Usability; Acceptability
Keywords: decision making for incapacitated patients; intensive care; surrogate decision making; patient centered care; Palliative Care; End of Life; Quality of Communication; Anxiety; Depression
MeSH Terms: conditions — Death; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSDM Tool (Experimental): Surrogate will complete educational sessions on CSDM tool prior to each family meeting with clinical team.
  Interventions: Other: CSDM Web-Based Tool Intervention
- Control (No Intervention): Surrogates will receive augmented usual care. The augmentation is that there will be 2 family meetings scheduled during the first 10 days of enrollment.

INTERVENTIONS:
Other: CSDM Web-Based Tool Intervention — The web and tablet-based tool is designed to help family members become familiar with ICU environment, routines, and clinicians, prepare for family meetings, and learn how to make values-based decisions for their loved one. The tool contains short videos, interactive exercises, and links to other resources. Family members work through the tool shortly after admission to the ICU, before each family meeting, and any other time they wish to during the ICU admission.
  Arms: CSDM Tool

SUMMARY:
The goal is to develop a pragmatic, scalable intervention to overcome problems with surrogate decision making in ICUs.

The aim is to conduct a pilot study among surrogates and clinicians of 50 incapacitated patients at high risk of death to assess the feasibility of deploying the web-based tool as well as to examine the tools impact on the patient and family outcome measures summarized in the hypotheses below.

DETAILED DESCRIPTION:
Roughly 600,000 Americans annually die in or shortly after an ICU admission, generally after decisions by surrogates to forego life support. Several decades of research indicate:

1. Family members in ICUs often struggle in the role of surrogate and experience high rates of lasting psychological sequelae (e.g. depression, anxiety, PTSD). For example, a systematic review found that one third of surrogates have long term feelings of guilt and doubt about the decisions they made.
2. Patients often receive treatment that is inconsistent with their values and preferences. For example, in the SUPPORT trial, physicians were frequently unaware of patients' wishes regarding end-of-life care, and patients often died receiving more invasive treatment than they preferred.
3. Intensive care near the end of life is a significant contributor to health care costs. For example, medical care in the last year of life accounts for 25% of Medicare costs, and ICU care contributes substantially.

Breakdowns in clinician-family communication in ICUs are common and an important target for interventions. Using quantitative analysis of audiorecorded goals of care discussions in ICUs, we found that in more than 50% of conversations clinicians did not inquire about the patient's values and treatment preferences, and in a similar proportion failed to explicitly offer alternatives to indefinite life-prolonging treatment, such as time-limited trials or comfort-focused treatment. We have also documented frequent omissions of important prognostic information during such conversations and other researchers have documented that surrogates often hold unduly optimistic estimates of patients' prognosis. These data highlight the importance of improving the quality of collaborative decision making in ICUs.

This proposal is responsive to national research priorities: The proposed research addresses priority areas for national action from the Institute of Medicine and NIH: improving clinician-family communication and end-of-life care for patients with advanced organ system failure. It is responsive to calls by the Institute on Aging to promote patient-centered decision making for elderly patients.

A critical barrier to addressing these problems is the absence of a scalable intervention. No empirically validated decision support tools exist for the range of critical illnesses confronted in ICUs. Prior interventions to address these problems (e.g., proactive palliative care consultation or adding a family support counselor to the ICU team) face major barriers to dissemination due to projected palliative care workforce shortages and the high cost of adding more personnel to ICU care teams.

A pragmatic, scalable intervention to overcome these problems has been developed. This pilot study among surrogates and clinicians of 50 incapacitated patients will assess the feasibility of deploying the web-based tool as well as to examine the tools impact on measures of communication and decision quality.

ELIGIBILITY:
Inclusion Criteria:

* Surrogate decision maker for ICU patient that lacks decisional capacity
* Permission from Patient's ICU Primary Attending Physician

Exclusion Criteria:

* Non-English Speaking
* Inability to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Intervention compliance | Duration of ICU stay, an expected average of 4 weeks
  Data tracking analytics will be employed to determine the extent to which the tool is used as per protocol.

SECONDARY OUTCOMES:
Participants' ratings of usability of the tool | Duration of hospital stay, an expected average of 4 weeks
  Usability of the tool will be measured with the System Usability Scale
Participants' ratings of acceptability of the tool | Duration of hospital stay, an expected average of 4 weeks
  Acceptability will be measured with the user Acceptability Assessment
Participants' ratings of perceived usefulness of the tool | Duration of hospital stay, an expected average of 4 weeks
  Usefulness will be measured with the Usefulness Assessment
Feasibility of enrolling family members in a critical care setting | Through study completion, estimate one year past primary start date
  Measured by meeting target enrollment
Feasibility of retaining family members in a critical care setting in a trial | Three months post-discharge
  The number of subjects that complete the long term follow up

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | Three months post-discharge
  To assess surrogate emotional state during intervention
Impact of Events Scale | Three months post-discharge
  To assess risk of post-traumatic stress disorder
Inventory of Complicated Grief | Three months post-discharge
  To assess complicated grief
Quality of Communication Scale | Three months post-discharge
  To assess communication between surrogates and clinicians
Mortality | Three months post-discharge
  Death
Functional status | Three months post-discharge
  To assess basic activities of daily living
Patient-Perceived Centeredness of Care Scale | Three months post-discharge
  To assess patient centeredness of care adapted for use by surrogates
Hospital costs | Three months post-discharge
  To assess costs of hospital
3-month health care utilization | Three months post-discharge
  To assess health care utilization over specified period

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B White, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Background] Azoulay E, Chevret S, Leleu G, Pochard F, Barboteu M, Adrie C, Canoui P, Le Gall JR, Schlemmer B. Half the families of intensive care unit patients experience inadequate communication with physicians. Crit Care Med. 2000 Aug;28(8):3044-9. doi: 10.1097/00003246-200008000-00061. PMID 10966293
- [Background] Lynn J, Teno JM, Phillips RS, Wu AW, Desbiens N, Harrold J, Claessens MT, Wenger N, Kreling B, Connors AF Jr. Perceptions by family members of the dying experience of older and seriously ill patients. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Ann Intern Med. 1997 Jan 15;126(2):97-106. doi: 10.7326/0003-4819-126-2-199701150-00001. PMID 9005760
- [Background] Schenker Y, Tiver GA, Hong SY, White DB. Association between physicians' beliefs and the option of comfort care for critically ill patients. Intensive Care Med. 2012 Oct;38(10):1607-15. doi: 10.1007/s00134-012-2671-4. Epub 2012 Aug 11. PMID 22885651
- [Background] Schenker Y, Tiver GA, Hong SY, White DB. Discussion of treatment trials in intensive care. J Crit Care. 2013 Oct;28(5):862-9. doi: 10.1016/j.jcrc.2013.04.015. Epub 2013 Jun 13. PMID 23768446
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] White DB, Braddock CH 3rd, Bereknyei S, Curtis JR. Toward shared decision making at the end of life in intensive care units: opportunities for improvement. Arch Intern Med. 2007 Mar 12;167(5):461-7. doi: 10.1001/archinte.167.5.461. PMID 17353493
- [Background] White DB, Engelberg RA, Wenrich MD, Lo B, Curtis JR. Prognostication during physician-family discussions about limiting life support in intensive care units. Crit Care Med. 2007 Feb;35(2):442-8. doi: 10.1097/01.CCM.0000254723.28270.14. PMID 17205000
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Wendler D, Rid A. Systematic review: the effect on surrogates of making treatment decisions for others. Ann Intern Med. 2011 Mar 1;154(5):336-46. doi: 10.7326/0003-4819-154-5-201103010-00008. PMID 21357911
- [Background] Riley GF, Lubitz JD. Long-term trends in Medicare payments in the last year of life. Health Serv Res. 2010 Apr;45(2):565-76. doi: 10.1111/j.1475-6773.2010.01082.x. Epub 2010 Feb 9. PMID 20148984
- [Background] Hogan C, Lunney J, Gabel J, Lynn J. Medicare beneficiaries' costs of care in the last year of life. Health Aff (Millwood). 2001 Jul-Aug;20(4):188-95. doi: 10.1377/hlthaff.20.4.188. PMID 11463076
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Prendergast TJ, Claessens MT, Luce JM. A national survey of end-of-life care for critically ill patients. Am J Respir Crit Care Med. 1998 Oct;158(4):1163-7. doi: 10.1164/ajrccm.158.4.9801108. PMID 9769276
- [Background] Fried TR, Bradley EH, Towle VR, Allore H. Understanding the treatment preferences of seriously ill patients. N Engl J Med. 2002 Apr 4;346(14):1061-6. doi: 10.1056/NEJMsa012528. PMID 11932474
- [Background] Sudore RL, Fried TR. Redefining the "planning" in advance care planning: preparing for end-of-life decision making. Ann Intern Med. 2010 Aug 17;153(4):256-61. doi: 10.7326/0003-4819-153-4-201008170-00008. PMID 20713793
- [Background] Hua MS, Li G, Blinderman CD, Wunsch H. Estimates of the need for palliative care consultation across united states intensive care units using a trigger-based model. Am J Respir Crit Care Med. 2014 Feb 15;189(4):428-36. doi: 10.1164/rccm.201307-1229OC. PMID 24261961
- [Background] Lupu D; American Academy of Hospice and Palliative Medicine Workforce Task Force. Estimate of current hospice and palliative medicine physician workforce shortage. J Pain Symptom Manage. 2010 Dec;40(6):899-911. doi: 10.1016/j.jpainsymman.2010.07.004. PMID 21145468
- [Background] O'Connor AM, Llewellyn-Thomas HA, Flood AB. Modifying unwarranted variations in health care: shared decision making using patient decision aids. Health Aff (Millwood). 2004;Suppl Variation:VAR63-72. doi: 10.1377/hlthaff.var.63. PMID 15471770
- [Background] O'Connor AM, Rostom A, Fiset V, Tetroe J, Entwistle V, Llewellyn-Thomas H, Holmes-Rovner M, Barry M, Jones J. Decision aids for patients facing health treatment or screening decisions: systematic review. BMJ. 1999 Sep 18;319(7212):731-4. doi: 10.1136/bmj.319.7212.731. PMID 10487995
- [Background] Stacey D, Bennett CL, Barry MJ, Col NF, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Legare F, Thomson R. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD001431. doi: 10.1002/14651858.CD001431.pub3. PMID 21975733